CLINICAL TRIAL: NCT03234855
Title: Laparoscopic Measuring Device Usability Study
Brief Title: Laparoscopic Measuring Device Study
Acronym: LMD-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Boehringer Labs LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: LMD-1
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Physician Feedback

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- LMD: Physician uses LMD during procedure.
  Interventions: Device: LMD

INTERVENTIONS:
Device: LMD — Physician uses LMD to measure defect during procedure.

SUMMARY:
This study is gathering opinions from surgeons on the usability of our laparoscopic measuring device.

DETAILED DESCRIPTION:
In June of 2016, SAGES (Society of American Gastrointestinal and Endoscopic Surgeons) issued a recommendation stating that:

"Surgeons should measure and document the size of the hernia defect they are repairing. The total area encompassing all the defects should be measured, and surgeons should be familiar with internal and external measurement techniques for all hernia locations, as well as how to avoid common measurement errors."

An incorrect mesh size can have detrimental consequences to the effectiveness of the mesh. According to the SAGES recommendation:

"Overestimating the defect size will result in the choice of a larger prosthetic size, which may be more difficult to handle and may have more laxity, allowing it to bulge into the defect more than if it was placed taut. The difficulty in prosthetic handling may also lead to errors in fixation, and the prosthetic can more easily sway between fixation points, due to the larger dimensions."

While a smaller mesh size can also be problematic:

"Underestimating the defect size may lead to choosing a prosthetic that is too small, thus increasing the risk of hernia recurrence." In order to aid surgeons in more accurately measuring hernia defects, Boehringer Labs LLC has developed a laparoscopic surgical measuring device. This study aims to obtain feedback from surgeons on the usefulness and design of the device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hernia defect that requires laparoscopic measurement

Exclusion Criteria:

* Minors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients whose physician has already decided that laparoscopic hernia repair surgery is the best route of treatment for a hernia defect.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Physician Feedback | 6 months
  Physician forms opinion on usefulness and design of LMD

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No patient data will be collected